CLINICAL TRIAL: NCT02220036
Title: Effect of Magnesium Supplementation on Kidney Function, Insulin Resistance and Metabolic Profile in Patients With Diabetic Nephropathy
Brief Title: Effect of Magnesium Supplementation on Patients With Diabetic Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Effect of Magnesium Supplementation on Kidney Function, Insulin Resistance and Metabolic Profile in Patients With Diabetic Nephropathy, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 198476
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes
Keywords: Diabetic nephropathy; Renal function; Insulin resistance; Metabolic profile; Serum magnesium level
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies; Insulin Resistance | interventions — Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium Oxide (Active Comparator): magnesium tablets, 250 milligram magnesium, 12 weeks, every day 1 tablet
  Interventions: Dietary Supplement: Magnesium Oxide
- Placebo (Placebo Comparator): Placebo tablets, the same in color, odor and appearance with magnesium tablets, 12 weeks, one tablet every day

INTERVENTIONS:
Dietary Supplement: Magnesium Oxide — Patients aged more than 18 years old with diabetic nephropathy having Fasting Blood Sugar more than 126 mg/dL and proteinuria 30-300 mg/dL (microalbuminuria) and Glomerular Filtration Rate more than 90 mL/min will be chosen. Patient group will receive magnesium supplement (250 milligram) and the other group will receive placebo which is similar to the magnesium tablets in color, odor and appearance both for 12 weeks. All subjects will complete 4 physical activity and 4 dietary records. Outcome measurements including metabolic, renal and inflammatory profiles will be measured at the beginning and end of the study as well as anthropometric measurements.
  Other Names: 21 Century company
  Arms: Magnesium Oxide

SUMMARY:
This is a double-blind randomized clinical trial which will start at June 2014 and end on June 2015 in Isfahan city. Serum creatinine level is considered as a key variable and the sample size calculated 80 persons (40 persons for control group and 40 persons for patient group). Patients aged more than 18 years old with diabetic nephropathy having Fasting Blood Sugar more than 126 mg/dL and proteinuria 30-300 mg/dL (microalbuminuria) and Glomerular Filtration Rate more than 90 mL/min will be chosen. Patient group will receive magnesium supplement (250 milligram) and the other group will receive placebo which is similar to the magnesium tablets in color, odor and appearance both for 12 weeks. All subjects will complete 4 physical activity and 4 dietary records. Outcome measurements including metabolic, renal and inflammatory profiles will be measured at the beginning and end of the study as well as anthropometric measurements.

DETAILED DESCRIPTION:
This is a double-blind randomized clinical trial which will start at June 2014 and end on June 2015 in Isfahan city. Serum creatinine level is considered as a key variable and the sample size calculated 80 persons (40 persons for control group and 40 persons for patient group).

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* diabetic nephropathy
* Fasting Blood Sugar more than 126 milligram per deciliter
* Proteinuria 30-300 milligram per deciliter (microalbuminuria)
* Glomerular Filtration Rate more than 90 milliliter per minute
* Not having hyperthyroidism or hypothyroidism
* Not having any feverish urinary tract infection
* Not using any kind of drug including Cigarette
* Not having any liver disease
* Not having any cancer and inflammatory diseases
* Not having more than 4 kilogram weight loss during last 3 months
* Not using any magnesium-rich supplement

Exclusion Criteria:

* changing medicine dose
* Not having adherence (using less than 75 percent of medicines)
* Cardiac Arrhythmias

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine | 12 weeks

SECONDARY OUTCOMES:
Blood Urine Nitrogen | 12 weeks
Glomerular Filtration Rate | 12 weeks
Proteinuria | 12 weeks
Fasting Blood Sugar | 12 weeks
Hemoglobin A1c | 12 weeks
Serum insulin level | 12 weeks
High Density Lipoprotein | 12 weeks
Low Density Lipoprotein | 12 weeks
Very Low Density Lipoprotein | 12 weeks
Triglyceride | 12 weeks
Total Cholesterol | 12 weeks
high sensitive C-Reactive Protein | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Sadeghian, Professor, Study Chair — Isfahan University of Medical Sciences
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran